CLINICAL TRIAL: NCT02505789
Title: Transfusion-related Epstein-Barr Virus (EBV) Infection Among Allogeneic Stem Cell Transplant Pediatric Recipients: a Multicenter Prospective Cohort Study (TREASuRE Study)
Brief Title: Transfusion-related EBV Infection Among Allogeneic Stem Cell Transplant Pediatric Recipients
Acronym: TREASuRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Blood Services (Other)
Responsible Party: Principal Investigator, Helen Trottier, Associate Professor, St. Justine's Hospital
Other Study IDs: CBS/CIHR_201209-293922
Record Dates: First submitted 2015-07-15; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Lymphoproliferative Disorders
Keywords: Epstein-Barr Virus; Post-transplant lymphoproliferative disease (PTLD); Infection; Cell Transplants; Herpesvirus 4, Human
MeSH Terms: conditions — Lymphoproliferative Disorders; Epstein-Barr Virus Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Determining the source of EBV in severe EBV infections — Blood units administered to patients with severe EBV infection will be traced back to the donors who in turn (with consent) will be serologically assessed for EBV, and all seropositive donors will have their EBV strain genotyped for comparison to the patient's strain.

SUMMARY:
In many countries, numerous steps are taken to minimize the risk of infection from transfused blood products. Typically, blood banking organisations will screen for an array of infectious pathogens as part of their quality control protocol. While transmission of these tested agents via transfusion has become exceedingly rare, the risk of transfusion-transmitted infections for which testing is not currently performed continues to be a concern. Among these untested infectious agents is Epstein-Barr virus (EBV, also known as human herpesvirus-4). Most notably, infection with this virus in transplant recipients can give rise to a malignant disorder called post-transplant lymphoproliferative disease (PTLD), a life-threatening complication which is due to the uncontrolled expansion of EBV-infected cells. It is also associated with other complications such as hepatitis, hemophagocytic syndrome, etc. in transplant population. It is recognised that EBV infection can occurred in transfused immune suppressed graft recipients but the origin of the viral infection is still a matter of debate. It is a known fact that the EBV already present in the recipient's blood can undergo reactivation due to immune suppression. However, because it is known to occur more frequently in patients who are EBV-seronegative at the time of transplant, it is also accepted that primary infection contracted via an infected graft can be a source of virus. The question we are seeking to answer is whether immune suppressed graft recipients can acquire primary EBV infection via transfusion of blood products. EBV is present in the blood of most adults and cases of EBV transfusion-related infection have been reported. Transplant populations are generally transfused with very large volumes of blood products and our recent pilot study supports the possibility that transfusion-related EBV infection can be transmitted to pediatric hematopoietic stem cell (HSCT) recipients (Trottier et al, 2012). The aim of this study is to analyse the risk of EBV transmission through blood product transfusion in pediatric allogeneic HSCT patients.

DETAILED DESCRIPTION:
All patients will be recruited approximately 1 month before transplantation (before pre-transplant conditioning chemotherapy and pre-surgery evaluation) and followed-up to 1 year post-transplantation. Thus, each subject will be followed-up for a 13-month period. At entry, a questionnaire will document socio-demographic data and pre-transplant clinical indicators such as age, gender, primary diagnosis, previous chemotherapy, previous transfusion, etc. During follow-up, case report forms (CRF) will allow prospective reporting of all variables pertaining to EBV serology, transplantation, blood product transfusion and EBV complication.

EBV PCR and serology testing:

This study is observational and will use the results of EBV PCR and EBV serology allowing our objectives to be achieved with considerable cost reduction. Time zero is when the patient receives his graft. Some tests are done before time zero (pre-transplant array of test including EBV serology). After time zero, in all sites, there is a follow-up treatment protocol including EBV PCR testing. Pre-transplant sera from recipients and donors are tested by standard methods for mmunoglobulin G (IgG) antibodies to the EBV capsid antigen (VCA), IgG antibodies to EBV early antigens (EA) and anticomplement antibodies to the EBV nuclear antigens (EBNA). EBV DNA testing is performed by quantitative polymerase chain reaction (PCR). Each centre has an established threshold value for determining viral load. In order to properly interpret the patients' viral load data from each participating center, all will be required to fill out a site report form (SRF) to describe their testing method for EBV PCR and EBV serology.

Pre-transplant measurement of EBV antibodies:

Serology testing, including EBV seroprevalence, is always done in all participating sites during the pre-transplant evaluation (before conditioning chemotherapy) in both donors and recipients. Serology testing is the test that is used to confirm the presence of the virus in the blood. For grafts provided by external sites, donor blood samples are always available and will allow for serology testing at the laboratory center where the transplantation is performed. Serology testing will not be done on cord-blood donor as it is virtually always negative for EBV. Donors and recipients will be classified according to their pre-transplant serology status as: 1) having past infection (VCA and EBNA IgG titers > 10), 2) having recent infection or being immune suppressed (VCA IgG titers > 10 and EBNA IgG titers < 10), 3) having reactivated infection (VCA, EBNA and EA IgG titers > 10), or 4) being naïve (no serological sign of prior infection).

Post-transplant EBV DNA PCR testing:

HSCT recipients are closely followed for EBV infection in the post-transplant period. Although most of the blood product transfusions occur during the peri-transplant period, it is possible that patients receive blood products at a later time post-transplantation. Follow-up on EBV PCR results and complications related to EBV will therefore continue up to one year post-transplant (or time of death). This time window will allow documentation of the entire clinical trajectory of HSCT. Protocols for follow-up after transplant, and for the diagnosis and treatment of EBV disease in allogeneic graft recipients have been reviewed in all participating sites. The incidence of EBV infection in recipients is measured by quantitative real-time PCR testing performed AT MINIMUM every 1-2 weeks from the time of transplant until hospital discharge (which is usually around 6 weeks post-transplantation). After hospital discharge, EBV PCR monitoring is performed at every clinical follow-up visit: AT LEAST twice per month for approximately 4-6 months post-transplant or as long as the patient remains immune suppressed. Thereafter, approximately one EBV PCR per month is performed until 1-year post-transplant.

In sum, the incidence of EBV infection will be adequately measured during a 1-year follow-up period. In all sites, AT LEAST 1 EBV PCR test is done per 1-2 weeks during hospitalization, 2 EBV PCR tests per month from hospital discharge to 6 months post-transplantation and approximately 1 EBV PCR test per month from 6 months to 12 months. The total number of EBV PCR results that will be collected per patient for the entire follow-up will be approximately 18. These results will be retrieved from patient charts.

PTLD and other complications related to EBV:

Clinical outcomes such as high and increasing viral load EBV infection and PTLD will be routinely screened until one year post-transplant. PTLD diagnosis will be made according to WHO criteria (Swerdlow et al, 2008) based on clinical or radiologic signs coexisting with an EBV-positive PCR on blood specimens. Information related to PTLD will be collected in the case report form. All other complications possibly related to EBV (for example: hemophagocytic syndrome, hepatitis, etc.) will also be documented. An adjudicating committee (C. Buteau and C Alfieri) will review patient-specific data elements to confirm PTLD and other complications related to EBV.

Transfused blood products:

Data on all blood products transfused will be collected and will include descriptors of the blood product unit (type of blood product, number of units, length of storage, etc.), volume transfused (milliliters), duration of the transfusion, as well as the date and time of each transfusion. Total volume received of every blood products will be considered in our analysis as well as the number of transfusions.

A site report form (SRF) will also be filled by each participating center to document its transfusion protocol such as the type of blood products used for HSCT, leukoreduction, type of red blood cells (RBCs) (washed, irradiated, CMV negative, etc.), type of plasma (fresh frozen plasma, frozen plasma, solvent detergent plasma), type of platelet concentrates (apheresis, pooled, etc,), maximum length of storage (days), etc.

Determining the source of EBV in severe EBV infections:

In order to demonstrate definitively that virus from transfused blood products can be linked to severe complications such as high and increasing viral load EBV infection/PTLD, we will genotype the EBV strain from these patients. Blood units administered to these patients will be traced back to the donors who in turn (with consent) will be serologically assessed for EBV, and all seropositive donors will have their EBV strain genotyped for comparison to the patient's strain. Many blood donors per case will have to be traced as recipients receive blood products from many blood donors (1 unit of RBC is provided by 1 donor, 1 unit of plasma is provided by 1 donor and 1 unit of platelet is provided by 4 donors). In average, we expected that about 25 donors will have to be traced per case (estimated with pilot data; Trottier et al, 2012). We are used in tracing blood donors of graft recipients as reported in Alfieri et al. (1996).

Brief procedure for EBV genotyping :

10 ml of blood (2 ml for infected pediatric patients) is separated by density centrifugation on Ficoll-hypaque gradients. The mononuclear cell fraction is harvested, washed and cultured in the presence of cyclosporine so as to allow outgrowth of the donor's EBV-positive cells and establishment of an immortalized EBV-positive B cell line. The viral DNA within this line can then be amplified by PCR using primers from the BamHI-K region of the EBV-genome, which is known to be highly polymorphic among the various EBV strains. The different sized fragments of the amplified region can be distinguished by migration on an agarose gel (Alfieri et al, 1996). In order to verify our results for identity between patients and blood donors we will also employ the EBNA-typing technique which is performed by western blot analysis using a defined EBNA-positive serum (Alfieri et al, 1996).

ELIGIBILITY:
Inclusion Criteria:

* patients receiving allogeneic HSCT (marrow, cord-blood, and peripheral blood stem cells)
* age below 21 years
* first HSCT

Exclusion Criteria:

-

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Only allogeneic HSCTs will be considered (no autologous grafts) because allogeneic grafts require a higher degree of immune suppression, which is known to increase risk with regard to EBV infection, development of PTLD and other EBV complications
Sampling Method: Non-Probability Sample
Enrollment: 324 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Measure of the risk of EBV infection in HSCT pediatric recipients from blood products transfusions (red blood cells, platelets, plasma) by EBV PCR and serology testing | 1 month before transplantation to 1 year post-transplantation
  EBV PCR and serology testing every 1-2 weeks until hospital discharge and at follow-up visit thereafter.

SECONDARY OUTCOMES:
Incidence of post-transplant EBV infection in allogeneic HSCT pediatric recipients stratified according to the EBV serostatus of the patient and the EBV status of the graft | 1 month before transplantation to 1 year post-transplantation
  Surveillance for PTLD and other EBV complications
Incidence of "high or increasing viral load EBV infection and PTLD" in allogeneic HSCT pediatric recipients stratified according to the EBV serostatus of the patient and the EBV status of the graft | 1 month before transplantation to 1 year post-transplantation
  Surveillance for PTLD and other EBV complications
Description of other complications related to EBV infection in this transplant population | 1 month before transplantation to 1 year post-transplantation
  Surveillance for PTLD and other EBV complications

CONTACTS AND LOCATIONS:
Overall Officials: Helen Trottier, PhD, Principal Investigator — St. Justine's Hospital
Locations (3):
- Canada (3):
  - BC Children's Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - St. Justine's Hospital, Montreal, Quebec

REFERENCES:
- [Background] Trottier H, Buteau C, Robitaille N, Duval M, Tucci M, Lacroix J, Alfieri C. Transfusion-related Epstein-Barr virus infection among stem cell transplant recipients: a retrospective cohort study in children. Transfusion. 2012 Dec;52(12):2653-63. doi: 10.1111/j.1537-2995.2012.03611.x. Epub 2012 Mar 15. PMID 22420319
- [Background] Alfieri C, Tanner J, Carpentier L, Perpete C, Savoie A, Paradis K, Delage G, Joncas J. Epstein-Barr virus transmission from a blood donor to an organ transplant recipient with recovery of the same virus strain from the recipient's blood and oropharynx. Blood. 1996 Jan 15;87(2):812-7. PMID 8555507